CLINICAL TRIAL: NCT04116281
Title: Study of the Possible Sensory, Biomechanical, Cardiorespiratory and Quality of Life Adaptations Associated With Physical Therapy Rehabilitation in the Short and Long Term Postoperative of Breast Cancer
Brief Title: Short and Long Term Effects of a Physical Therapy Program After Breast Cancer Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic situation
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Ivana Leão Ribeiro, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 154/2019
Record Dates: First submitted 2019-09-29; First posted 2019-10-04 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Upper limb function; Heart hate variability; Physical therapy; Breast neoplasms; Pressure pain threshold; Perceived pain
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised group (Experimental): Supervised group
  Interventions: Other: Rehabilitation after breast cancer surgery
- No supervised group (Other): Control group
  Interventions: Other: Rehabilitation after breast cancer surgery

INTERVENTIONS:
Other: Rehabilitation after breast cancer surgery — All participants are going to receive physical therapy intervention after breast cancer surgery at least removal drenaige. After that, will be randomized in two groups: Group 1 are going to receive a physical therapy program supervised by a physiotherapist; Group 2 are going to receive some instructions about the same program to perfomr at home without supervision. Both groups are going to receive 3 and 6 months of rehabilitation program.

SUMMARY:
Objectives: To evaluate the pressure pain threshold, shoulder biomechanics, cardiorespiratory function and the quality of life associated with the short and long-term physical therapy rehabilitation following breast cancer surgery. Methodology: The study presents three objectives and involves three groups of participants. Objective 1 is to develop a topographic map of pressure pain in the shoulder (using a digital pressure algometer), evaluate the biomechanics of the shoulder (using a digital inclinometer and load card), cardiorespiratory function (through frequency variability resting heart rate and distance traveled, through the six-minute walk test) and quality of life (through questionnaires of quality of life, anxiety, depression, sleep quality, upper limb functionality, fatigue and level of physical activity) between a group of women prior to the operation of breast cancer (experimental group, n = 36) and a group of asymptomatic controls for shoulder pain (control group, n = 18). Objective 2 is to evaluate the possible changes in the pain map over 24 weeks of supervised kinetic intervention (Supervised Physiotherapy experimental group, n = 18, will begin after drainage, frequency 3 times per week and duration of 60 minutes each session) compared to unsupervised kinetic intervention (Home Physiotherapy experimental group, n = 18, participants will receive an exercise booklet). Objective 3 is to evaluate the biomechanics of the shoulder, cardiorespiratory function and the quality of life with respect to the experimental group with and without kinesic supervision. To achieve objective 1, two baseline evaluations will be carried out in both experimental and control groups (considering the month prior to the surgery of the experimental group) and the average of the evaluations will be considered evaluation 1. To achieve objectives 2 and 3, evaluation 2 (after 4 weeks of intervention), 3 (after 12 weeks of intervention) and 4 (after 24 weeks of intervention) will be performed. The statistical analysis will include the examination of qualitative and quantitative variables. Statistical tests will be applied according to the normality of the data and a significance level of 5% will be adopted for all comparisons. Expected results: It is expected to identify sensory, biomechanical, cardiorespiratory and quality of life alterations in the experimental group, compared to the control group. In addition, after 24 weeks of intervention, the supervised experimental group will show improvement in all the aforementioned variables with respect to the unsupervised group.

ELIGIBILITY:
Inclusion Criteria:

* Surgical indication of conservative or removal breast surgery, associated with axillary lymphadenectomy or sentinel lymph node biopsy
* Any type of breast cancer
* Age range over 18 years

Exclusion Criteria:

* Breast cancer recurrence;
* Surgical treatment for bilateral breast cancer;
* Presence of lymphedema in the upper limb, measured by means of cirtometry of the upper limb with a measuring tape 14, asymmetries of more than 1.5 cm between the limbs were considered edema;
* Diagnosis of metastases;
* Shoulder pain compatible with shoulder compression symptoms as determined by the positive Hawkins-Kennedy test 30;
* Previous history of surgery and fractures in the upper extremities.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold over the shoulder of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to pressure pain threshold assessment over the shoulder at three and six monthes of treatment.
Pressure pain threshold over the shoulder of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to pressure pain threshold assessment over the shoulder at three and six monthes of treatment.
Strength grip of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to objective measurement that consist in to do a maximal strenth grip. The unity of measurement it is in kg.
Strength grip of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to objective measurement that consist in to do a maximal strenth grip. The unity of measurement it is in kg.

SECONDARY OUTCOMES:
Upper limb functionality of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to a questionnaire of upper limb function during activity daily routine. The questionnaire has 33 questions and each one has 5 posible answers.
Upper limb functionality of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to a questionnaire of upper limb function during activity daily routine. The questionnaire has 33 questions and each one has 5 posible answers.
Fatigue of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to a questionnaire wich contains 9 preguntas and 10 differente posibilities of answers.
Fatigue of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to a questionnaire wich contains 9 questions and 10 different posibilities of answers.
Cardiopulmonary function of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to functional capacity performed wiht the walking test measured by the distance performed after a walking.
Cardiopulmonary function of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to functional capacity performed wiht the walking test measured by the distance performed after a walking.
Cardiopulmonary function of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to heart rate variability measured with a Polar and reloj in a supine and orthostatic posture
Cardiopulmonary function of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to heart rate variability measured with a Polar and reloj in a supine and orthostatic posture
Quality of life of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Three months
  This outcome will involve data regarding to a questionnaire of quality of life regarding symptoms of chemotherapy that affects on quality of life perception. The questionnaire has 53 questions and each one has 4 posible answers.
Quality of life of breast cancer patients after a physical therapy rehabilitation program following the surgery. | Six months
  This outcome will involve data regarding to a questionnaire of quality of life regarding symptoms of chemotherapy that affects on quality of life perception. The questionnaire has 53 questions and each one has 4 posible answers.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana L Ribeiro, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Catholic University of Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Yes